CLINICAL TRIAL: NCT03580733
Title: Prospective Multicentre Randomized Double-blind Study Comparing Caspofungin to Placebo for the Treatment of ICU Intra-abdominal Candidiasis
Brief Title: Study Comparing Caspofungin to Placebo for the Treatment of ICU Intra-abdominal Candidiasis
Acronym: CASPER
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PI2018_843_0007
Record Dates: First submitted 2018-06-08; First posted 2018-07-09 (Actual); Last update posted 2024-07-10 (Actual); Status verified 2024-07

CONDITIONS: ICU Yeast Intra-abdominal Infection
Keywords: ICU; yeast intra abdominal infection; candidiasis; ß-D-glucan; caspofungin
MeSH Terms: conditions — Candidiasis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- placebo (Placebo Comparator): placebo
  Interventions: Other: placebo
- antifungal therapy (Experimental): caspofungin
  Interventions: Drug: caspofungin antifungal therapy

INTERVENTIONS:
Drug: caspofungin antifungal therapy — caspofungin
  Arms: antifungal therapy
Other: placebo — placebo
  Arms: placebo

SUMMARY:
The incidence of intra-abdominal candidiasis is increasing, and it is now the leading indication for antifungal therapy, ahead of candidemia. Prospective randomized trials of antifungal therapy have almost exclusively concerned patients with candidemia and did not include patients with intra-abdominal infections. The aim of this study is to demonstrate that caspofungin antifungal therapy for intra-abdominal candidiasis in ICU patients is associated with lower failure rate compared to placebo.

DETAILED DESCRIPTION:
The incidence of intra-abdominal candidiasis is increasing, and it is now the leading indication for antifungal therapy, ahead of candidemia. These infections are clearly associated with increased morbidity and mortality in both community-acquired and healthcare-associated infections. So far,prospective randomized trials of antifungal therapy have almost exclusively concerned patients with candidemia and did not include patients with intra-abdominal infections. No prospective randomized trial has been conducted on intra-abdominal candidiasis and most retrospective analyses have reported very conflicting results concerning the impact of treatment on outcome. The aim of this study is therefore to demonstrate that caspofungin antifungal therapy for intra-abdominal candidiasis in ICU patients is associated with lower failure rate compared to placebo.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years old
* Covered by national health insurance
* Admitted to ICU after surgery for intra-abdominal infection :

  * With suspected intra-abdominal candidiasis defined by a Peritonitis score ≥ 3(1)
  * Or with documented intra-abdominal candidiasis defined by positive direct examination or positive culture of peritoneal fluid collected intraoperatively.
* With written and signed informed consent

Exclusion Criteria:

* Allergy to caspofungin
* Life expectancy ≤ 48h
* Expected withdrawal of treatment
* Radiological drainage without surgery
* Severe hepatic impairment (Child-Pugh C score)
* Pregnant or lactating women
* Immunodepression (treatment including long-term corticosteroids, anti-TNF or disease including transplant patients)
* Infected acute pancreatitis
* Ascites fluid infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 448 (Estimated)
Dates: Start 2019-01-01 (Actual); Primary Completion 2024-10-04 (Estimated); Study Completion 2024-12-04 (Estimated)

PRIMARY OUTCOMES:
failure rate after the beginning of treatment | 28 days
  28-day failure rate after the beginning of treatment

SECONDARY OUTCOMES:
mortality | 28 and 90 days
  28 and 90-day mortality rate
success rate at the end of treatment | 8 days
  success rate at the end of treatment
slope of ß-D-glucan concentrations | 8 days
  slope of ß-D-glucan concentrations
mortality | 28 days
  28- 28 day mortality for subgroup analysis

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Amiens, Amiens, France

IPD SHARING:
Plan to Share IPD: No